CLINICAL TRIAL: NCT03148626
Title: Can a Mindfulness Curriculum Prevent Burnout During Pediatric Internship? A Multi-center Cluster Randomized Controlled Trial.
Brief Title: Does a Mindfulness Curriculum Prevent Physician Burnout During Pediatric Internship?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston Children's Hospital (Other); UCSF Benioff Children's Hospital Oakland (Other); Children's Hospital Medical Center, Cincinnati (Other); Floating Hospital for Children (Other); Nationwide Children's Hospital (Other); MaineHealth (Other); Saint Peters University Hospital (Other); University of California, Davis (Other); University of Florida (Other); University of Massachusetts, Worcester (Other); Seattle Children's Hospital (Other); Advocate Lutheran General Hospital (Other); University of Pittsburgh (Other); Loyola University Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-36221
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Burnout, Professional
Keywords: mindfulness curriculum
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Intervention Model Description: Multi-center cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINDI mindfulness curriculum (Experimental): The intervention is a seven-session mindfulness curriculum to be delivered over six months to pediatric interns.
  Interventions: Other: MINDI mindfulness curriculum
- Control (Placebo Comparator): Usual education.
  Interventions: Other: Control

INTERVENTIONS:
Other: MINDI mindfulness curriculum — A seven-session mindfulness curriculum implemented over six-months during pediatric internship.
  Arms: MINDI mindfulness curriculum
Other: Control — Usual Education
  Arms: Control

SUMMARY:
A triad of exhaustion, depersonalization and inefficacy, physician burnout is an epidemic among trainees associated with delivering poor quality care. Training programs are desperate for evidence-based programs that can prevent burnout during residency. Mindfulness training programs can reduce burnout among primary care physicians, but have not been tested during physician training. Pilot testing of a novel mindfulness curriculum during pediatric internship was found to be feasible to implement.

The primary objective of this study is to determine if implementing a novel 6-month mindfulness curriculum comprised of seven 1-hour sessions can reduce physician burnout and increase mindfulness practice and empathy. A multicenter cluster randomized controlled trial will be conducted among interns training in programs of various sizes and regions to address this objective. The investigators hypothesize that completing a mindfulness curriculum during internship will reduce interns' levels of physician burnout and increase their mindfulness practice and empathy.

Within pairs in pediatric residency programs matched on size (a proxy for burnout), clusters of interns in each program will be randomized to experience either the mindfulness curriculum over a 6-month period (intervention) or receive the usual educational curriculum (control). During a 15-month study period, burnout, mindfulness and empathy will be assessed using validated measures at baseline, 6- and 15-month follow-up. The impact of the intervention will be determined by comparing physician burnout, empathy and mindfulness scores between interns in the intervention and control groups. This methodologically rigorous multi-center cluster RCT will determine if implementing an innovative 6-month mindfulness curriculum reduces pediatric interns' burnout and improves empathy and mindfulness practice.

DETAILED DESCRIPTION:
Rationale and Purpose: The unacceptably high prevalence of burnout during residency has made training programs desperate for evidence-based programs designed to prevent burnout during residency. Mindfulness training programs have been shown to reduce burnout and depression among primary care physicians as well as in a myriad of other professions. The investigators' longitudinal pilot test of implementing an innovative mindfulness curriculum in a large busy pediatric internship was determined to be feasible and acceptable. However, the absence of a control group, small sample size, and single residency program site limited the detection of meaningful statistically significant differences in levels of burnout, mindfulness, or empathy that could have generalizable value.

Study Objectives: A methodologically rigorous study will be conducted to determine if a 6-month mindfulness curriculum implemented during pediatric internship can reduce physician burnout and increase mindfulness practice and empathy. The investigators hypothesize that completing a mindfulness curriculum during internship will reduce interns' levels of physician burnout and increase their mindfulness practice and empathy.

Outcome Measures: The primary outcome measure will be physician burnout, assessed by the emotional-exhaustion sub-scale of Maslach Burnout Inventory (MBI). Many studies use this sub-scale as the sole measure of burnout because "emotional-exhaustion is considered the most central aspect of burnout." Secondary outcomes will include: burnout as a dichotomous measure, defined as emotional exhaustion scores >=27 or depersonalization scores >=10, per MBI guidelines; participants' levels of mindfulness, based on the Five Facet Mindfulness Questionnaire; and empathy, assessed by the Jefferson Scale of Physician Empathy. These measures were selected based on prior conceptual frameworks and the model of factors related to burnout.

Study Design: A large multi-center, stratified, cluster, randomized, controlled trial of the 7-session mindfulness curriculum in pediatric residency programs will be implemented and analyzed. To ensure that interns training in the same program have the same educational experience, clustered randomization will be conducted centrally using a computer-generated random allocation sequence. After pairing pediatric residency programs based on size as a proxy for baseline burnout, the clusters of interns in each program will be randomized to experience either: 1) the enhanced mindfulness curriculum over a 6-month period or 2) usual educational curriculum (control). Control group subjects will be blinded to knowing what the intervention group received, but the intervention subjects will not be blinded to participating in the mindfulness sessions.

Study Intervention: Programs randomized to the intervention arm will be asked to deliver the mindfulness curriculum to interns over their first 6 months of training (from July through December of the academic year)following the MINDI facilitator guide, which includes facilitator preparation materials, frequently asked questions, and detailed instructions for running the seven sessions of the mindfulness curriculum. . The lack of a robust impact on mindfulness practice in the previous pilot implementation of the MINDI curriculum suggests that hour-long mindfulness sessions delivered once a month over 6 months may not be a frequent enough intervention to change interns' behavior. Thus, the investigators will enhance the intervention by including 10 minutes of guided meditation at the start of regularly scheduled clinical didactic sessions (e.g. noontime conference) two weeks after each of the 7 MINDI sessions. Programs randomized to the control arm will not change their current curriculum but will be given the facilitator guide after the study is completed.

Study Procedures: Subjects in the intervention arm will experience the seven-session mindfulness curriculum over a 6-month period. These sessions will be delivered during the routine didactic schedule that the residency program uses to educate their interns (e.g. noon conferences and/or weekly educational afternoons, etc). Subjects in the Control arm will receive the usual educational curriculum. The investigators will assess independent and dependent measures by inviting subjects to complete voluntary, de-identified surveys three times duringthe one-year study period: at baseline (before the 1st MINDI session, which may be given during intern orientation), and at 6-months and then 15-months after course initiation. Non-investigator staff will offer a modest incentive to subjects who return completed surveys to maximize the completion rates.

Statistical Methods: The numbers and rates of physician burnout, and the mean, median, and range of the scores for mindfulness, empathy, and the emotional-exhaustion sub-scale of burnout will be calculated. Bivariate comparisons will be done between these outcome measures and selected demographic measures. Comparisons between the control and intervention groups will be performed using chi-square tests for dichotomous outcomes (such as burnout) and t-tests for continuous measures. Multivariate clustered logistic and linear regressions analysis will be conducted to determine independent predictors of dichotomous outcomes and continuous measures, while controlling for randomization group assignment and dependent measures associated with the outcomes. the size of clusters in the study to vary since cluster randomization of nequal numbers of subjects typically produces uneven group-sizes. All unadjusted and adjusted regressions will be clustered on residency program.

ELIGIBILITY:
Inclusion Criteria: All members of the intern class (e.g. post-graduate year 1) of pediatric residency programs who enrolled in this study will be eligible to participate in this study.

Exclusion Criteria: None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change in physician burnout from baseline to 6-month follow-up | Will be measured at baseline and 6-month follow-up
  Physician burnout will be measured using the Maslach Burnout Inventory.
Change in physician burnout from baseline to 15-month follow-up | Will be measured at baseline and 15-month follow-up
  Physician burnout will be measured with the Maslach Burnout Inventory.

SECONDARY OUTCOMES:
Change in empathy from baseline to 6 mo follow-up | Will be measured at baseline and both 6-month follow-up
  Empathy will be measured using the Jefferson Scale of Physician Empathy and/or Davis's Interpersonal Reactivity Index.
Change in empathy from baseline to 15 mo follow-up | Will be measured at baseline and 6-month follow-up
  Empathy will be measured using the Jefferson Scale of Physician Empathy and/or Davis's Interpersonal Reactivity Index.
Change in mindfulness from baseline to 6 mo follow-up | Will be measured at baseline and 15-month follow-up
  Mindfulness, a mental state achieved by focusing one's awareness on the present moment while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations, will be measured using the Five Facet Mindfulness Questionnaire.
Change in mindfulness from baseline to 15 mo follow-up | Will be measured at baseline and 15-month follow-up
  Mindfulness, a mental state achieved by focusing one's awareness on the present moment while calmly acknowledging and accepting one's feelings, thoughts, and bodily sensations, will be measured using the Five Facet Mindfulness Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Sox, MD, MS, Study Director — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraiman YS, Cheston CC, Cabral HJ, Allen C, Asnes AG, Barrett JT, Batra M, Bernstein W, Bleeker T, Dietz PM, Lewis J, Li ST, Ma TM, Mahan JD, Michelson CD, Poynter SE, Vining MA, Watson K, Sox CM. Effect of a Novel Mindfulness Curriculum on Burnout During Pediatric Internship: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Apr 1;176(4):365-372. doi: 10.1001/jamapediatrics.2021.5740. PMID 35072694